CLINICAL TRIAL: NCT02404194
Title: Optimizing Cognitive Training to Improve Functional Outcome in Clinical High Risk (CHR)
Brief Title: Targeted Cognitive Training in Clinical High Risk (CHR) for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Beth Israel Deaconess Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christine Hooker, Professor, Department of Psychiatry and Behavioral Sciences, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH105246; R01MH105246 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Clinical High Risk for Psychosis
Keywords: schizophrenia; psychosis; at risk; prodrome; attenuated psychosis syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Cognitive Training (Experimental): 40 hours of computerized cognitive training
  Interventions: Behavioral: Targeted Cognitive Training
- Computer Games (Placebo Comparator): 40 hours of computer games
  Interventions: Behavioral: Computer Games

INTERVENTIONS:
Behavioral: Targeted Cognitive Training — Targeted Cognitive Training is performed on the computer through Posit Science. Games are modern and engaging modifications of classic neuropsychological tests, such as set-shifting games modeled on the Wisconsin Card Sort Test, and cognitive control games modeled on Stroop-like interference tasks. Games will target two sets of skills: Targeted cognitive skills include: processing speed, memory, attention, flexibility/cognitive-control, and problem-solving. After 20 hours of training on these skills, participants will complete 20 hours of training on core social cognitive skills, including facial affect recognition, gaze direction perception, and face identity recognition, and theory of mind.
  Other Names: Posit Science
  Arms: Targeted Cognitive Training
Behavioral: Computer Games — The comparison intervention consists of 40 hours of commercially available and cognitively non-specific computer games. These computer games - such as checkers, solitaire, crossword puzzles - are entertaining and engaging but do not target specific neurocognitive skills.
  Arms: Computer Games

SUMMARY:
This project is a randomized-controlled trial to test the efficacy of computer-based targeted cognitive training (TCT) versus a placebo intervention of commercial computer games in adolescent/young adults at clinical high risk (CHR) for psychosis. TCT is designed to optimize learning-induced neuroplasticity in vulnerable neurocognitive systems. A main aim is to test the hypothesis that this neuroscience-guided TCT intervention will improve neural function, and that these neural improvements will improve cognition and functional outcome. CHR participants will be randomly assigned to 40 hours of TCT or placebo computer games completed within 10 weeks. TCT consists of 20 hours of training in cognition, including processing speed, memory, attention, and cognitive control followed by 20 hours of training in social cognition including affect recognition and theory of mind. Neuroimaging, cognition, social cognition, clinical symptoms, and functional status will be assessed at baseline, after 20 hours/5 weeks of cognitive training (mid-intervention), and after 20 hours/5 weeks of social-cognitive training (post-intervention). Cognition, social cognition, symptoms, and functioning will also be assessed at a 9 month follow-up (i.e. 9 months after intervention completion). We predict that TCT will lead to improvements in neurocognitive function and functional status. The results of this study will provide important information about a benign, non-pharmacological intervention for improving cognition and functional outcome in CHR individuals.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* One or more psychosis-risk syndromes as defined by the Structured Interview for Psychosis-Risk Syndromes (SIPS)

Exclusion Criteria:

* Intelligence Quotient (IQ) < 70
* Major medical illness or neurological disorder
* Lifetime history of Axis I psychotic disorder and/or clear evidence that psychosis-risk syndrome is due to non-schizophrenia-spectrum Axis I or Axis II disorder

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2015-03; Primary Completion 2020-11-23 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery | Change in cognition from baseline (pre-intervention) to 10 weeks (post-intervention)
  Behavioral assessment of cognition

SECONDARY OUTCOMES:
Global Function: Social and Role Scales | Change in functioning from baseline (pre-intervention) to 10 weeks (post-intervention)
  Behavioral assessment of daily functioning

CONTACTS AND LOCATIONS:
Overall Officials: Christine I Hooker, PhD, Principal Investigator — Rush University Medical Center, Dept of Psychiatry & Behavioral Sciences
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- See also: Website for Dr. Hooker's Laboratory — http://scholar.harvard.edu/chooker/home